CLINICAL TRIAL: NCT05478980
Title: The Effects of a Multi-ingredient Night-time Tea on Sleep Quality, Wellbeing and Markers of Immune Function: a Randomised, Controlled, Crossover Study
Brief Title: The Effects of a Multi-ingredient Night-time Tea on Sleep Quality, Wellbeing and Markers of Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 50CE1
Record Dates: First submitted 2021-10-27; First posted 2022-07-28 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2021-10

CONDITIONS: Mood; Poor Quality Sleep; Good Sleep Habit; Sleep
Keywords: Sleep; Mood; Physical health; Mental health; Immunological function
MeSH Terms: conditions — Sleep Hygiene; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Tea - Good Sleepers (Experimental)
  Interventions: Dietary Supplement: Night Time Tea
- Control Tea - Good Sleepers (Active Comparator)
  Interventions: Dietary Supplement: Control Tea
- Active Tea - Poor Sleepers (Experimental)
  Interventions: Dietary Supplement: Night Time Tea
- Control Tea - Poor Sleepers (Active Comparator)
  Interventions: Dietary Supplement: Control Tea

INTERVENTIONS:
Dietary Supplement: Night Time Tea — Night-time Tea
  Arms: Active Tea - Good Sleepers; Active Tea - Poor Sleepers
Dietary Supplement: Control Tea — Feel New Tea
  Arms: Control Tea - Good Sleepers; Control Tea - Poor Sleepers

SUMMARY:
The aim of the study is to determine whether a night-time tea can improve subjective sleep quality in healthy sleepers and self-reported poor sleepers, compared to a control drink.

DETAILED DESCRIPTION:
The study will adopt a randomised, double-blind, placebo controlled, crossover design. Sixty-eight healthy adults aged 18+ (34 good sleepers and 34 poor sleepers) will be recruited from the general population. Good sleepers will be recruited if they have a stable sleep-wake schedule (i.e. bed/wake time within the range of 22.00 - 09.00 and with at least 6.5 hours of sleep duration reported per night). Poor sleepers will be recruited if they report subjective sleep difficulties (i.e. poor sleep quality or unrefreshing sleep) and if they display a Pittsburgh Sleep Quality Index total score of >5. Participants will consume both an active tea, and a control tea in a counterbalanced order for 7 days (separated by a 7-day washout period). Participants will complete questionnaires assessing mood, quality of life and sleep and provide blood samples to assess immunological markers. Sleep monitoring will also be conducted using actigraphy sleep monitoring and sleep diaries. Assessments will be made at baseline and following 7 days supplementation.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female adults aged 18 years and above. Both good sleepers and poor sleepers will be recruited. Good sleepers will be recruited if they have a stable sleep-wake schedule (i.e. bed/wake time within the range of 22.00 - 09.00 and with at least 6.5 hours of sleep duration reported per night).

Poor sleepers will be recruited if they report subjective sleep difficulties (i.e. poor sleep quality or unrefreshing sleep) and if they display a Pittsburgh Sleep Quality Index total score of >5.

Exclusion Criteria:

Both good and poor sleeper participants cannot participate if they display evidence of current or previous sleep disorders (e.g. sleep apnoea, insomnia, circadian rhythm disorders); an initial screening for sleep disorders will be conducted using the Sleep Disorders Screening Checklist - 25 (SDS-CL).

* Participants must not be shift workers
* Cannot currently be participating in other research trials which will compromise the results here
* Participants cannot take part if they will be sleeping at a location other than their usual residence during participation
* Nor if they have experienced travel across multiple time zones within the last three months or will be experiencing travel across multiple time zones during the study
* Participants cannot take part if they have current or previous mood disturbances
* Are currently unwell with anything that impacts sleep
* Are currently using medication which affects the central nervous system
* Or are currently misusing alcohol or drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Consensus sleep diary (CSD) - Subjective sleep quality | Following 7 days of intervention

SECONDARY OUTCOMES:
Consensus sleep diary (CSD) - Subjective sleep continuity (Total sleep time) | Following 7 days of intervention
Consensus sleep diary (CSD) - Subjective sleep continuity (Time in bed) | Following 7 days of intervention
Consensus sleep diary (CSD) - Subjective sleep continuity (Sleep efficiency %) | Following 7 days of intervention
Consensus sleep diary (CSD) - Subjective sleep continuity (Sleep latency) | Following 7 days of intervention
Consensus sleep diary (CSD) - Subjective sleep continuity (Number of awakenings and wake after sleep onset) | Following 7 days of intervention
Karolinska Sleepiness Scale (KSS) | Following 7 days of intervention
Positive and negative affect schedule (PANAS) | Following 7 days of intervention
World Health Organization Quality of Life- Brief (WHOQOL-BREF) | Following 7 days of intervention
Short-Form Health Survey 36 (SF-36) | Following 7 days of intervention
Actigraphy objective sleep measures (Time in bed) | Following 7 days of intervention
Actigraphy objective sleep measures (Total sleep time) | Following 7 days of intervention
Actigraphy objective sleep measures (Sleep efficiency %) | Following 7 days of intervention
Actigraphy objective sleep measures (Number of awakenings) | Following 7 days of intervention
Actigraphy objective sleep measures (Sleep latency) | Following 7 days of intervention
Actigraphy objective sleep measures (wake after sleep onset) | Following 7 days of intervention
Immunological markers (Interleukins-6) | Following 7 days of intervention
Immunological markers (Interleukins-10) | Following 7 days of intervention
Immunological markers (Tumour Necrosis Factor - alpha (TNF-a)) | Following 7 days of intervention
Immunological markers (C-Reactive protein) | Following 7 days of intervention
Immunological markers (Cortisol) | Following 7 days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Dodd, Principal Investigator — Northumbria University
Locations (1):
- Brain Performance Nutrition Research Centre, Newcastle upon Tyne, Tyne & Wear, United Kingdom